CLINICAL TRIAL: NCT00587236
Title: A Blinded Comparison of Conventional Colonoscopy to Endoscopic AFI and NBI for Dysplasia Detection in Patients With Ulcerative Colitis and Sclerosing Cholangitis or Known Colorectal Dysplasia or Cancer- A Pilot Clinical Study
Brief Title: Compare Conventional Colonosocpy to Endoscopic AFI, NBI for Dysplasia Detection for Ulcerative Colitis & Cholangitis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher J. Gostout, PI, Mayo Clinic
Other Study IDs: 5-06
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Colitis, Ulcerative; Cholangitis, Sclerosing
Keywords: Autofluorescence; Narrow Band; High definition white light
MeSH Terms: conditions — Colitis, Ulcerative; Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with chronic ulcerative colitis and concurrent primary sclerosing cholangitis.
- 2: Patients with chronic ulcerative colitis and known dysplasia or cancer.

SUMMARY:
This study is being done to:

To attempt to increase the detection of precancerous colon tissue in patients with chronic ulcerative colitis and primary sclerosing cholangitis;

To determine if an investigational scope that can look at the lining of the colon in different ways will help the doctor identify abnormal tissue in patients with chronic ulcerative colitis and concurrent primary sclerosing cholangitis; and

To determine if this investigational scope can accurately detect precancerous or cancerous tissue in patients with chronic ulcerative colitis that are known to have had cancerous or precancerous tissue in the past.

DETAILED DESCRIPTION:
Patients with concurrent chronic ulcerative colitis and primary sclerosing cholangitis or patients with chronic ulcerative colitis and known colorectal dysplasia or cancer, presenting for surveillance colonoscopy will be recruited. After giving informed consent patients will then undergo colonoscopy in a segmental fashion. Colonoscopy with white light will be performed to the cecum and examination will be performed on withdrawal. First conventional white light will be used to examine the cecum and ascending colon and random biopsies will be obtained. All endoscopically apparent lesions will be biopsied separately. Immediately following will be examination of that segment of cecum and ascending colon under AFI first, then NBI with targeted biopsies of suspicious areas being taken. The AFI and NBI modality will be achieved by simply flipping a switch.. If necessary, washing of oozing blood from random biopsy sites will be performed., The remainder of the colon will be assessed in like fashion: transverse, descending and rectosigmoid. Because high definition endoscopy is the default modality, this will be in use throughout the procedure.

All lesions detected will be documented and biopsied for a maximum of four biopsies per suspicious lesion. Note will be taken of which modality resulted in visualization of the lesion. Data on the factors under study will be collected: i) disease type (CUC + PSC or CUC with known dysplasia), ii) Age, iii) Sex, iv) length of time with disease, v) extent of disease, vi) the interaction between iv and v will be collected. In addition, dysplasia yes/no will be established after biopsy histology is established and the modality under which abnormalities were observed will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring a clinically indicated surveillance colonoscopy
* able to give informed written consent
* history of chronic ulcerative colitis and colonic dysplasia/or cancer or primary sclerosing cholangitis

Exclusion Criteria:

* patients with known colonic obstruction
* INR ./= 2.5 or thrombocytopenia ,50,000
* patients with clinically important cardiopulmonary disease who are unable to safely undergo prolonged conscious sedation
* pregnancy
* symptomatic coronary artery disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with chronic ulcerative colitis and Primary sclerosing cholangitis and/or patients with chronic ulcerative colitis and known colorectal dysplasia or cancer needing a surveillance colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2006-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Compare the dysplasia detection rate between scope modalities and biopsy type; surveillance or targeted biopsies in CUC patients with concurrent PSC. | Two years

SECONDARY OUTCOMES:
Assess the impact of patient related factors on the difference in dysplasia detection rate between while light colonoscopy and the AFI and NBI techniques in patients with CUC and concurrent PSC. | Two years.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Gostout, MD, Study Director — Mayo Clinic, Rochester, MN
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Eaden JA, Abrams KR, Mayberry JF. The risk of colorectal cancer in ulcerative colitis: a meta-analysis. Gut. 2001 Apr;48(4):526-35. doi: 10.1136/gut.48.4.526. PMID 11247898
- [Background] Provenzale D, Onken J. Surveillance issues in inflammatory bowel disease: ulcerative colitis. J Clin Gastroenterol. 2001 Feb;32(2):99-105. doi: 10.1097/00004836-200102000-00003. PMID 11205664
- [Background] Kornbluth Am J Gastroenterology 2004 Practice Guidelines for UC in adults as an additional reference
- [Background] Rubin CE, Haggitt RC, Burmer GC, Brentnall TA, Stevens AC, Levine DS, Dean PJ, Kimmey M, Perera DR, Rabinovitch PS. DNA aneuploidy in colonic biopsies predicts future development of dysplasia in ulcerative colitis. Gastroenterology. 1992 Nov;103(5):1611-20. doi: 10.1016/0016-5085(92)91185-7. PMID 1426881
- [Background] Taylor BA, Pemberton JH, Carpenter HA, Levin KE, Schroeder KW, Welling DR, Spencer MP, Zinsmeister AR. Dysplasia in chronic ulcerative colitis: implications for colonoscopic surveillance. Dis Colon Rectum. 1992 Oct;35(10):950-6. doi: 10.1007/BF02253497. PMID 1395982
- [Background] Rembacken BJ, Fujii T, Cairns A, Dixon MF, Yoshida S, Chalmers DM, Axon AT. Flat and depressed colonic neoplasms: a prospective study of 1000 colonoscopies in the UK. Lancet. 2000 Apr 8;355(9211):1211-4. doi: 10.1016/s0140-6736(00)02086-9. PMID 10770302
- [Background] Kudo S, Tamura S, Nakajima T, Yamano H, Kusaka H, Watanabe H. Diagnosis of colorectal tumorous lesions by magnifying endoscopy. Gastrointest Endosc. 1996 Jul;44(1):8-14. doi: 10.1016/s0016-5107(96)70222-5. PMID 8836710
- [Background] Kiesslich R, Fritsch J, Holtmann M, Koehler HH, Stolte M, Kanzler S, Nafe B, Jung M, Galle PR, Neurath MF. Methylene blue-aided chromoendoscopy for the detection of intraepithelial neoplasia and colon cancer in ulcerative colitis. Gastroenterology. 2003 Apr;124(4):880-8. doi: 10.1053/gast.2003.50146. PMID 12671882
- [Background] Rutter MD, Saunders BP, Schofield G, Forbes A, Price AB, Talbot IC. Pancolonic indigo carmine dye spraying for the detection of dysplasia in ulcerative colitis. Gut. 2004 Feb;53(2):256-60. doi: 10.1136/gut.2003.016386. PMID 14724160
- [Background] Kara MA, Peters FP, Ten Kate FJ, Van Deventer SJ, Fockens P, Bergman JJ. Endoscopic video autofluorescence imaging may improve the detection of early neoplasia in patients with Barrett's esophagus. Gastrointest Endosc. 2005 May;61(6):679-85. doi: 10.1016/s0016-5107(04)02577-5. PMID 15855971
- [Background] Haringsma J, Tytgat GN. The value of fluorescence techniques in gastrointestinal endoscopy: better than the endoscopist's eye? I: The European experience. Endoscopy. 1998 May;30(4):416-8. doi: 10.1055/s-2007-1001292. No abstract available. PMID 9689518
- [Background] Nakayoshi T, Tajiri H, Matsuda K, Kaise M, Ikegami M, Sasaki H. Magnifying endoscopy combined with narrow band imaging system for early gastric cancer: correlation of vascular pattern with histopathology (including video). Endoscopy. 2004 Dec;36(12):1080-4. doi: 10.1055/s-2004-825961. PMID 15578298
- [Background] Hamamoto Y, Endo T, Nosho K, Arimura Y, Sato M, Imai K. Usefulness of narrow-band imaging endoscopy for diagnosis of Barrett's esophagus. J Gastroenterol. 2004 Jan;39(1):14-20. doi: 10.1007/s00535-003-1239-z. PMID 14767729
- [Background] Machida H, Sano Y, Hamamoto Y, Muto M, Kozu T, Tajiri H, Yoshida S. Narrow-band imaging in the diagnosis of colorectal mucosal lesions: a pilot study. Endoscopy. 2004 Dec;36(12):1094-8. doi: 10.1055/s-2004-826040. PMID 15578301
- [Background] Toruner M, Harewood GC, Loftus EV Jr, Sandborn WJ, Tremaine WJ, Faubion WA, Schroeder KW, Egan LJ. Endoscopic factors in the diagnosis of colorectal dysplasia in chronic inflammatory bowel disease. Inflamm Bowel Dis. 2005 May;11(5):428-34. doi: 10.1097/01.mib.0000158951.54388.3a. PMID 15867581
- [Background] Lachin JM. Introduction to sample size determination and power analysis for clinical trials. Control Clin Trials. 1981 Jun;2(2):93-113. doi: 10.1016/0197-2456(81)90001-5. PMID 7273794
- [Background] Riddell RH, Goldman H, Ransohoff DF, Appelman HD, Fenoglio CM, Haggitt RC, Ahren C, Correa P, Hamilton SR, Morson BC, et al. Dysplasia in inflammatory bowel disease: standardized classification with provisional clinical applications. Hum Pathol. 1983 Nov;14(11):931-68. doi: 10.1016/s0046-8177(83)80175-0. PMID 6629368